CLINICAL TRIAL: NCT01526733
Title: A Phase 4, Randomized, Double-Blind, 2-Way Crossover Study of Continuous Subcutaneous Insulin Infusion (CSII) With, Compared to Without, Pretreatment With Recombinant Human Hyaluronidase (rHuPH20)
Brief Title: Randomized, Double Blind, 2 Way Crossover Study of CSII With, Versus Without, Pretreatment With Human Hyaluronidase
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Halo-117-401
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; Continuous Subcutaneous Insulin Infusion (CSII)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — salicylhydroxamic acid; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin (Aspart or Lispro)-Sham (Sham Comparator): In Phase I or Phase II of the study, participants received 0.15 units per kilogram (U/kg) insulin (either insulin aspart or insulin lispro) as a continuous subcutaneous insulin infusion (CSII) for 16 days, with sham injections administered prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16.
  Each Phase was separated by a washout period of 5 to 21 days.
  Interventions: Drug: Sham Injection; Drug: Insulin aspart; Drug: Insulin lispro
- Insulin (Aspart or Lispro)-rHuPH20 (Experimental): In Phase I or Phase II of the study, participants received 0.15 U/kg insulin (either insulin aspart or insulin lispro) as a CSII for 16 days. Prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16, participants received a 1 mL (150 U) injection of recombinant human hyaluronidase (rHuPH20).
  Each Phase was separated by a washout period of 5 to 21 days.
  Interventions: Drug: Recombinant human hyaluronidase PH20; Drug: Insulin aspart; Drug: Insulin lispro

INTERVENTIONS:
Drug: Sham Injection
  Arms: Insulin (Aspart or Lispro)-Sham
Drug: Recombinant human hyaluronidase PH20
  Other Names: rHuPH20; PH20; Hylenex
  Arms: Insulin (Aspart or Lispro)-rHuPH20
Drug: Insulin aspart
  Other Names: Novolog; Aspart
Drug: Insulin lispro
  Other Names: Humalog; Lispro

SUMMARY:
The purpose of this study is to evaluate consistency of accelerated insulin absorption and onset-of-action and shortened duration of action for bolus insulin infusions after pretreatment with 150 units (U) of Hylenex® (recombinant human hyaluronidase PH20 [rHuPH20]) injection at the time of infusion set insertion compared to sham injection.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of age 18 to 65 years, inclusive. Females of child-bearing potential must use a standard and effective means of birth control for the duration of the study.
2. Non-smoking participants with Type 1 diabetes mellitus (T1DM) treated with insulin for ≥12 months. Nonsmoking means abstinence from cigarettes and cigars for 3 months and negative cotinine screening tests at screening.
3. Body mass index (BMI) 18.0 to 35.0 kilograms per meter squared (kg/m²), inclusive.
4. Glycosylated hemoglobin A1c (HbA1c) ≤10% based on local laboratory results.
5. Fasting connecting peptide of insulin (C-peptide) <0.6 nanograms per milliliter (ng/mL).
6. Current treatment with insulin <90 units per day (U/d).
7. Current use of rapid acting insulin analog.
8. Routine use of CSII as the primary route of insulin administration for at least 3 months prior to screening
9. Participants should be in good general health based on medical history and physical examination without medical conditions that might prevent the completion of study drug infusions and assessments required in the study protocol.

Exclusion Criteria:

1. Known or suspected allergy to any component of any of the study drugs in this study.
2. Previous enrollment in this study.
3. Use of drugs that may interfere with the interpretation of study results or are known to cause clinically relevant interference with insulin action, glucose utilization, or recovery from hypoglycemia. Participants taking maintenance doses of blood thinners (for example, coumadin or heparin) will be excluded.
4. Use of any long-acting insulin injection within 72 hours of Study Day 1; participants will continue to refrain from use throughout the duration of the study (Phases I and II).
5. Recurrent major hypoglycemia or hypoglycemic unawareness, as judged by the Investigator.
6. Current addiction to alcohol or substances of abuse as determined by the Investigator.
7. Blood donation or phlebotomy (>500 milliliters [mL]) within the previous 8 weeks of the Screening Visit(s) in this study.
8. Pregnancy, breastfeeding, the intention of becoming pregnant, or not using adequate contraceptive measures (adequate contraceptive measures consist of sterilization, intra-uterine device [IUD], oral or injectable contraceptives, or barrier methods).
9. Symptomatic gastroparesis.
10. Receipt of any investigational drug within 4 weeks of Study Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States

REFERENCES:
- See also: Sponsor's Website — http://www.halozyme.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin-rHuPH20, Then Insulin-sham: In Phase I, participants received 0.15 units per kilogram (U/kg) insulin (either insulin aspart or insulin lispro) as a continuous subcutaneous insulin infusion (CSII) for 16 days. Prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16, participants received a 1 milliliter (mL) (150 U) injection of recombinant human hyaluronidase PH20 (rHuPH20).
  In Phase II, participants received 0.15 U/kg insulin (either insulin aspart or insulin lispro) as a CSII for 16 days, with a sham injections administered prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16.
  Phase I and II were separated by a washout period of 5 to 21 days.
- Insulin-sham, Then Insulin-rHuPH20: In Phase I, participants received 0.15 U/kg insulin (either insulin aspart or insulin lispro) as a CSII for 16 days, with a sham injection administered prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16.
  In Phase II, participants received 0.15 U/kg insulin (either insulin aspart or insulin lispro) as a CSII for 16 days. Prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16, participants received a 1 mL (150 U) injection of rHuPH20.
  Phase I and Phase II were separated by a washout period of 5 to 21 days.
Period: Phase 1
Arm/Group | Insulin-rHuPH20, Then Insulin-sham | Insulin-sham, Then Insulin-rHuPH20
Started | 12 | 13 (One participant discontinued after receiving insulin-sham and before receiving insulin-rHuPH20.)
Received at Least 1 Dose of Study Drug | 12 | 13
Completed | 10 | 12
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: Washout Period of 5 to 21 Days
Arm/Group | Insulin-rHuPH20, Then Insulin-sham | Insulin-sham, Then Insulin-rHuPH20
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0
Period: Phase 2
Arm/Group | Insulin-rHuPH20, Then Insulin-sham | Insulin-sham, Then Insulin-rHuPH20
Started | 10 | 12
Completed | 10 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Enrolled Participants: All participants enrolled in the study.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Early Insulin Exposure (%AUC[0-60])
Description: Early insulin exposure, defined as the percentage of total insulin exposure (area under the insulin concentration curve [AUC{0 360}]) that occurs within the first hour following bolus dose of insulin during the 2 euglycemic clamps is presented. Blood samples were collected 10 minutes predose and at 0, 5, 10, 15, 20, 30, 45, and 60 minutes postdose during a euglycemic clamp.
Time Frame: 10 minutes predose; 0, 5, 10, 15, 20, 30, 45, and 60 minutes postdose on Days 1 and 4
Population: Participants who completed both phases of the study and with evaluable %AUC(0-60) data.
Measure: Mean (Standard Deviation); unit: percentage of AUC(0-60)
Groups:
- Insulin (Aspart or Lispro)-rHuPH20: In Phase I or Phase II of the study, participants received 0.15 U/kg insulin (either insulin aspart or insulin lispro) as a CSII for 16 days. Prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16, participants received a 1 mL (150 U) injection of rHuPH20.
  Each Phase was separated by a washout period of 5 to 21 days.
- Insulin (Aspart or Lispro)-Sham: In Phase I or Phase II of the study, participants received 0.15 U/kg insulin (either insulin aspart or insulin lispro) as a CSII for 16 days, with sham injections administered prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16.
  Each Phase was separated by a washout period of 5 to 21 days.
Arm/Group | Insulin (Aspart or Lispro)-rHuPH20 | Insulin (Aspart or Lispro)-Sham
Number analyzed (Participants) | 21 | 21
percentage of AUC(0-60)
  Day 1 | 33.53 (11.81) | 17.85 (8.24)
  Day 4 | 39.45 (9.72) | 33.52 (10.78)
Statistical Analysis 1: Comparison: Insulin (Aspart or Lispro)-rHuPH20 vs Insulin (Aspart or Lispro)-Sham; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Comparison of Day 1 Insulin (Aspart or Lispro)-rHuPH20 versus Day 1 Insulin-sham; A mixed model with fixed effects for treatment, day, and interaction of treatment with day was performed using a compound symmetric covariance matrix; Geometric Least Squares Mean Ratio = 2.15, 90% CI 2-sided [1.71 to 2.71]
Statistical Analysis 2: Comparison: Insulin (Aspart or Lispro)-rHuPH20 vs Insulin (Aspart or Lispro)-Sham; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Comparison of Day 4 Insulin (Aspart or Lispro)-rHuPH20 versus Day 1 Insulin-sham; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares Mean Ratio = 2.62, 90% CI 2-sided [2.08 to 3.29]

2. Secondary Outcome: Maximum Glucose Infusion Rate (GIRmax)
Description: Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose on Days 1 and 4
Population: Participants who completed both phases of the study and with evaluable GIRmax data.
Measure: Mean (Standard Deviation); unit: milligrams/kilogram/minute
Arm/Group | Insulin (Aspart or Lispro)-rHuPH20 | Insulin (Aspart or Lispro)-Sham
Number analyzed (Participants) | 21 | 21
milligrams/kilogram/minute
  Day 1 | 13.47 (5.46) | 11.14 (4.21)
  Day 4 | 10.75 (3.73) | 11.83 (3.26)

3. Secondary Outcome: Time to First Occurrence of Maximum Glucose Infusion Rate (tGIRmax)
Description: as for outcome 2
Time Frame: 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose on Days 1 and 4
Population: Participants who completed both phases of the study and with evaluable tGIRmax data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Insulin (Aspart or Lispro)-rHuPH20 | Insulin (Aspart or Lispro)-Sham
Number analyzed (Participants) | 21 | 21
minutes
  Day 1 | 78.95 (37.16) | 132.62 (55.07)
  Day 4 | 81.86 (45.99) | 97.38 (47.31)

4. Secondary Outcome: Time to 50% Maximum Glucose Infusion Rate (tGIR50%Max)
Description: Early and late tGIR50%max are presented. Blood samples were collected at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose on Days 1 and 4
Population: Participants who completed both phases of the study and with evaluable early and late tGIR50%max data.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Insulin (Aspart or Lispro)-rHuPH20 | Insulin (Aspart or Lispro)-Sham
Number analyzed (Participants) | 21 | 21
minutes
  Early tGIR50%, Day 1 | 40.33 (20.13) | 54.67 (33.97)
  Late tGIR50%, Day 1 | 114.52 (54.33) | 152.14 (61.00)
  Early tGIR50%, Day 4 | 32.57 (14.50) | 39.67 (15.51)
  Late tGIR50%, Day 4 | 113.24 (48.72) | 126.71 (50.37)

5. Secondary Outcome: Time to 50% Total Glucose Infused (50%Gtot)
Description: as for outcome 2
Time Frame: 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose on Days 1 and 4
Population: Participants who completed both phases of the study and with evaluable 50%Gtot data.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Insulin (Aspart or Lispro)-rHuPH20: In Phase I or Phase II of the study, participants received 0.15 U/kg insulin (either insulin aspart or insulin lispro) as a CSII for 16 days. Prior to outpatient euglycemic clamps on Days 1 and 4 and prior to outpatient meal test procedures on Days 7, 10, 13, and 16, participants received a 1 mL (150 U) rHuPH20.
  Each Phase was separated by a washout period of 5 to 21 days.
Arm/Group | Insulin (Aspart or Lispro)-rHuPH20 | Insulin (Aspart or Lispro)-Sham
Number analyzed (Participants) | 21 | 21
minutes
  Day 1 | 40.33 (20.13) | 32.57 (14.50)
  Day 4 | 54.67 (54.67) | 39.67 (15.51)

6. Secondary Outcome: Area Under the Glucose Concentration Curve (AUC[0-360])
Description: Area under the glucose concentration curve from 0 to 360 minutes (AUC[0-360]) is presented. Blood samples were collected 30 and 10 minutes prior to insulin bolus and at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 30 minutes and 10 minutes predose; 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose on Days 1 and 4
Population: Participants who completed both phases of the study and with evaluable AUC(0-360) data.
Measure: Mean (Standard Deviation); unit: picomoles*minutes/liter
Arm/Group | Insulin (Aspart or Lispro)-rHuPH20 | Insulin (Aspart or Lispro)-Sham
Number analyzed (Participants) | 21 | 21
picomoles*minutes/liter
  Day 1 | 1312.41 (627.33) | 1199.54 (535.80)
  Day 4 | 1063.77 (500.06) | 1139.65 (414.94)

7. Secondary Outcome: Duration of Insulin Action (AUMC[0-360]/AUC[0-360])
Description: Duration of insulin action was calculated by dividing the area under the first moment curve (AUMC[0-360]) by the area under the concentration versus time curve (AUC[0-360]). AUCM is the total area under the first moment curve. First moment curve is obtained by plotting concentration-time versus time. It can be used to measure how long a drug stays in the body. Blood samples were collected 10 minutes predose and at 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose during a euglycemic clamp.
Time Frame: 10 minutes predose; 0, 5, 10, 15, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, and 360 minutes postdose on Days 1 and 4
Population: Participants who completed both phases of the study and with evaluable AUMC(0-360)/AUC(0-360) data.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Insulin (Aspart or Lispro)-rHuPH20 | Insulin (Aspart or Lispro)-Sham
Number analyzed (Participants) | 21 | 21
ratio
  Day 1 | 119.02 (21.18) | 154.03 (27.58)
  Day 4 | 111.25 (20.59) | 120.57 (20.85)

ADVERSE EVENTS:
Description: Insulin was not considered a study drug for safety assessments and causality assessments were done for rHuPH20 only.
Arm/Group | Insulin (Aspart or Lispro)-rHuPH20 | Insulin (Aspart or Lispro)-Sham
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 13/24 | 9/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin (Aspart or Lispro)-rHuPH20 (N=24) | Insulin (Aspart or Lispro)-Sham (N=23)
Anaemia (Blood and lymphatic system disorders) | 2 | 4
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Injection site pain (General disorders) | 3 | 1
Injection site pruritus (General disorders) | 1 | 2
Injection site haemorrhage (General disorders) | 1 | 0
Injection site haematoma (General disorders) | 1 | 0
Injection site induration (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 0 | 1
Tenderness (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information obtained as a result of this study or during the conduct of this study will be regarded as confidential. The Investigator agrees to use the information for the purpose of carrying out this study and for no other purpose, unless prior written permission from the Sponsor (Halozyme) is obtained.